CLINICAL TRIAL: NCT06280300
Title: Intensive Multi-Disciplinary Care Initiative for Patients With Newly Diagnosed Brain Metastases
Brief Title: Multi-disciplinary Care for Brain Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Alissa Thomas, Associate Professor of Neurological Sciences, University of Vermont Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UVMMC2203
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Brain Metastases, Adult
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Other: health services intervention
- Multidisciplinary Care (Experimental)
  Interventions: Other: health services intervention

INTERVENTIONS:
Other: health services intervention — Health services intervention

SUMMARY:
This is a health services intervention study aimed at understanding the impact of intensive multi-disciplinary care compared with standard care on patient-reported symptom outcomes and prognostic awareness in patients with brain metastases.

DETAILED DESCRIPTION:
This is a cohort study of patient with newly diagnosed brain metastases assigned to standard of care (SOC) or intensive multi-disciplinary care (IMDC). Care for all patients with brain metastases involves complex medical decision making and requires input for multiple stakeholders, including medical oncology, neurosurgery, radiation oncology, and neuro-oncology. Palliative care should be an essential component of the care team for all patients with brain metastases by the very nature of this advanced malignancy. At the University of Vermont, our current process for diagnosis and management of patients with brain metastases relies heavily on the physician and team who make the initial diagnosis to consult others as they see appropriate. This process may look different for different patients. We rationalize that a systematic approach with intensive multidisciplinary care (IMDC) will benefit patients with brain metastases by providing consistent access to multi-disciplinary discussion.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all genders must be at least 18 years of age.
* Patients must have histologically confirmed, newly diagnosed brain metastases from known or suspected solid tumor primary neoplasms.
* Patients must be able to accurately provide self-report data (e.g. per clinical judgment, cognitive function is intact).
* Patients must be able to complete questionnaires in English.
* Patients must have the ability to provide informed consent.

Exclusion Criteria:

* Patients who are < 18 years of age are not eligible.
* Patients who are Pregnant are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient reported outcomes | 6-12 months
  Symptom burden based on patient reporting on Brain Mets Symptom Inventory

SECONDARY OUTCOMES:
Feasibility | 6-12 months
  Number of % of patients able to complete protocol-specified activities
Patient understanding of prognosis | 6-12 months
  Concordance with physician predication of prognosis
survival | 6-12 months
  Survival outcomes for patients receiving best supportive care

OTHER OUTCOMES:
Exploratory survival outcome | 6-12 months
  90 day and 1 year survival

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No